CLINICAL TRIAL: NCT02326298
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Group, Study Followed by a Dose-Blind Period and Open-Label Follow-Up to Evaluate the Efficacy and Safety of Certolizumab Pegol in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: An Efficacy and Safety Study of Two Dose Levels of Certolizumab Pegol (CZP) in Subjects With Plaque Psoriasis (PSO)
Acronym: CIMPASI-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0005; 2014-003513-28 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2014-12-22; First posted 2014-12-29 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Psoriasis; Plaque Psoriasis
Keywords: Certolizumab Pegol; Cimzia; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CZP 200 mg (Experimental): CZP 400 mg at Weeks 0, 2, 4, followed by CZP 200 mg every two weeks (Q2W) from Week 6 to Week 14.
  Treatment received from Week 16-48 is based on initial treatment and response to treatment:
  * PASI50 responders at Week 16 continue to receive CZP 200 mg Q2W.
  * PASI50 non-responders at Week 16 will be removed from blinded study medication and escape to unblinded CZP 400 mg Q2W. Subjects who receive unblinded CZP 400 mg Q2W for 16 weeks and do not achieve a PASI50 response will be withdrawn from the study.
  * PASI50 non-responders at Week 32 or a later time point will be withdrawn from the study.
  Subjects who complete the Maintenance Period (with PASI50 response at Week 48) enter the Open-label Extension Period on CZP 200 mg Q2W.
  Week 48 completers in the escape arm continue to receive CZP 400 mg Q2W or may switch to CZP 200 mg Q2W.
  Depending on PASI50 or PASI75 responses at Week 60 or a later time point, subjects may switch to CZP 400 mg Q2W or withdraw from the study.
  Interventions: Biological: Certolizumab Pegol
- CZP 400 mg (Experimental): CZP 400 mg every two weeks (Q2W) through Week 14.
  Treatment received from Week 16 - 48 is based on initial treatment and response to treatment:
  * PASI50 responders at Week 16 continue to receive CZP 400 mg Q2W.
  * PASI50 non-responders at Week 16 will be removed from blinded study medication and escape to CZP 400 mg Q2W. Subjects who receive unblinded CZP 400 mg Q2W for 16 weeks and do not achieve a PASI50 response will be withdrawn from the study.
  * PASI50 non-responders at Week 32 or a later time point will be withdrawn from the study.
  Subjects who complete the Maintenance Period (with PASI50 response at Week 48) enter the Open-label Extension (OLE) Period on CZP 200 mg Q2W. Week 48 completers in the escape arm continue to receive CZP 400 mg Q2W or may switch to CZP 200 mg Q2W.
  Subjects who achieve a PASI75 response during the OLE Phase may switch to CZP 200 mg Q2W.
  Interventions: Biological: Certolizumab Pegol
- Placebo (Placebo Comparator): Placebo subcutaneous (sc) injection every two weeks (Q2W).
  Treatment received from Week 16 - 48 is based on initial treatment and response to treatment:
  * PASI50 responders at Week 16, who do not achieve a PASI75 response at Week 16 receive CZP 400 mg at Weeks 16, 18 and 20 (loading doses) followed by CZP 200 mg Q2W starting at Week 22.
  * PASI75 responders at Week 16 continue to receive Placebo.
  * PASI50 non-responders at Week 16 will be removed from blinded study medication and escape to CZP 400 mg Q2W. Subjects who receive unblinded CZP 400 mg Q2W for 16 weeks and do not achieve a PASI50 response will be withdrawn from the study.
  * PASI50 non-responders at Week 32 or a later time point will be withdrawn from the study.
  Subjects who complete the Maintenance Period (with PASI50 response at Week 48) enter the Open-label Extension Period on CZP 200 mg Q2W. Week 48 completers in the escape arm continue to receive CZP 400 mg Q2W or may switch to CZP 200 mg Q2W.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Certolizumab Pegol — * Active Substance: Certolizumab Pegol
  * Pharmaceutical Form: Solution for injection in pre-filled syringe
  * Concentration: 200 mg/mL
  * Route of Administration: Subcutaneous use
  Other Names: Cimzia; CDP870; CZP
  Arms: CZP 200 mg; CZP 400 mg
Other: Placebo — * Active Substance: Placebo
  * Pharmaceutical Form: Solution for injection in pre-filled syringe
  * Concentration: 0.9 % saline
  * Route of Administration: Subcutaneous use
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of two dose levels of certolizumab pegol in adults with moderate to severe chronic plaque psoriasis when administered every 2 weeks.

DETAILED DESCRIPTION:
This study consists of the following Periods:

* Initial Treatment Period from Week 0 to Week 16
* Maintenance Treatment Period from Week 16 to Week 48
* Open-label Treatment Period from Week 48 to Week 144
* Safety Follow-Up Period from Week 144 to Week 152

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent
* Adult men or women >= 18 years
* Chronic plaque psoriasis for at least 6 months
* Baseline psoriasis activity and severity index >= 12 and body surface area >= 10 % and Physician's Global Assessments score >= 3
* Candidate for systemic psoriasis therapy and/or phototherapy and/or chemophototherapy
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Erythrodermic, guttate, generalized pustular form of psoriasis
* History of current, chronic, or recurrent infections of viral, bacterial, or fungal origin as described in the protocol
* Congestive heart failure
* History of a lymphoproliferative disorder including lymphoma or current signs and symptoms suggestive of lymphoproliferative disease
* Concurrent malignancy or a history of malignancy as described in the protocol
* History of, or suspected, demyelinating disease of the central nervous system (e.g., multiple sclerosis or optic neuritis)
* Female subjects who are breastfeeding, pregnant, or plan to become pregnant during the study or within 5 months following last dose of study drug (in Czech Republic and Germany) and within 3 months for all other countries. Male subjects who are planning a partner pregnancy during the study or within 10 weeks following the last dose of study drug
* Any other condition which, in the Investigator's judgment, would make the subject unsuitable for participation in the study
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2016-03-08 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (30):
- United States (8):
  - Ps0005 504, San Diego, California
  - Ps0005 502, West Des Moines, Iowa
  - Ps0005 500, Baton Rouge, Louisiana
  - Ps0005 506, Boston, Massachusetts
  - Ps0005 505, St Louis, Missouri
  - Ps0005 507, Albuquerque, New Mexico
  - Ps0005 508, Nashville, Tennessee
  - Ps0005 501, Houston, Texas
- Canada (7):
  - Ps0005 597, Edmonton, Alberta
  - Ps0005 591, Surrey, British Columbia
  - Ps0005 596, Ajax, Ontario
  - Ps0005 590, Hamilton, Ontario
  - Ps0005 593, Toronto, Ontario
  - Ps0005 595, Drummondville, Quebec
  - Ps0005 594, Québec, Quebec
- Czechia (4):
  - Ps0005 553, Náchod
  - Ps0005 550, Olomouc
  - Ps0005 551, Ostrava-Poruba
  - Ps0005 552, Prague
- Germany (8):
  - Ps0005 562, Mahlow, Brandenburg
  - Ps0005 565, Witten, North Rhine-Westphalia
  - Ps0005 569, Lübeck, Schleswig-Holstein
  - Ps0005 560, Berlin
  - Ps0005 561, Dresden
  - Ps0005 563, Hamburg
  - Ps0005 568, Hamburg
  - Ps0005 566, Kiel
- Hungary (3):
  - Ps0005 580, Orosháza, Bekes County
  - Ps0005 582, Budapest
  - Ps0005 581, Pécs

REFERENCES:
- [Result] Gottlieb AB, Blauvelt A, Thaci D, Leonardi CL, Poulin Y, Drew J, Peterson L, Arendt C, Burge D, Reich K. Certolizumab pegol for the treatment of chronic plaque psoriasis: Results through 48 weeks from 2 phase 3, multicenter, randomized, double-blinded, placebo-controlled studies (CIMPASI-1 and CIMPASI-2). J Am Acad Dermatol. 2018 Aug;79(2):302-314.e6. doi: 10.1016/j.jaad.2018.04.012. Epub 2018 Apr 13. PMID 29660421
- [Derived] Gisondi P, Gottlieb AB, Elewski B, Augustin M, McBride S, Tsai TF, de la Loge C, Fierens F, Lopez Pinto JM, Tilt N, Lebwohl M. Long-Term Health-Related Quality of Life in Patients with Plaque Psoriasis Treated with Certolizumab Pegol: Three-Year Results from Two Randomised Phase 3 Studies (CIMPASI-1 and CIMPASI-2). Dermatol Ther (Heidelb). 2023 Jan;13(1):315-328. doi: 10.1007/s13555-022-00861-4. Epub 2022 Dec 13. PMID 36509889
- [Derived] Gordon KB, Warren RB, Gottlieb AB, Blauvelt A, Thaci D, Leonardi C, Poulin Y, Boehnlein M, Brock F, Ecoffet C, Reich K. Long-term efficacy of certolizumab pegol for the treatment of plaque psoriasis: 3-year results from two randomized phase III trials (CIMPASI-1 and CIMPASI-2). Br J Dermatol. 2021 Apr;184(4):652-662. doi: 10.1111/bjd.19393. Epub 2020 Sep 9. PMID 32652544
- [Derived] Blauvelt A, Paul C, van de Kerkhof P, Warren RB, Gottlieb AB, Langley RG, Brock F, Arendt C, Boehnlein M, Lebwohl M, Reich K. Long-term safety of certolizumab pegol in plaque psoriasis: pooled analysis over 3 years from three phase III, randomized, placebo-controlled studies. Br J Dermatol. 2021 Apr;184(4):640-651. doi: 10.1111/bjd.19314. Epub 2020 Sep 6. PMID 32531798
- See also: Related Info — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in December 2014 and concluded in October 2018 from multiple sites in Europe and North America. 234 participants were included in the Randomized Set (RS) shown in the Participant Flow.
Pre-assignment Details: The study included a 5 Week Screening Period, a Double-blind Initial Treatment Period up to Week 16, a Dose-blind Maintenance Treatment Period up to Week 48, an Open-label Treatment Period up to Week 144 and a Post Study Safety Follow-up Period up to Week 152.
  Participant Flow refers to the Randomized Set, Open Label Set and Maintenance Set.
Groups:
- Placebo Q2W: Placebo sc injection Q2W.
  Treatment received from Week 16 - 48 was based on initial treatment and response to treatment:
  * PASI50 responders at Week 16, who did not achieve a PASI75 response at Week 16 received CZP 400 mg at Weeks 16, 18 and 20 (loading doses) followed by CZP 200 mg Q2W starting at Week 22.
  * PASI75 responders at Week 16 continued to receive Placebo.
  * PASI50 non-responders at Week 16 were removed from blinded study medication and escaped to unblinded CZP 400 mg Q2W. Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study.
  * PASI50 non-responders at Week 32 or a later time point were withdrawn from the study.
  Participants who completed the Maintenance Period (with PASI50 response at Week 48) entered the Open-label Extension (OLE) Period on CZP 200 mg Q2W. Week 48 completers in the escape arm continued to receive CZP 400 mg Q2W or may have switched to CZP 200 mg Q2W.
- CZP 200 mg Q2W: CZP 400 mg at Weeks 0, 2, 4, followed by CZP 200 mg Q2W from Week 6 to Week 14.
  Treatment received from Week 16 - 48 was based on initial treatment and response to treatment:
  * PASI50 responders at Week 16 continued to receive CZP 200 mg Q2W.
  * PASI50 non-responders at Week 16 were removed from blinded study medication and escaped to unblinded CZP 400 mg Q2W. Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study.
  * PASI50 non-responders at Week 32 or a later time point were withdrawn from the study.
  Participants who completed the Maintenance Period (with PASI50 response at Week 48) entered the OLE Period on CZP 200 mg Q2W.
  Week 48 completers in the escape arm continued to receive CZP 400 mg Q2W or may have switched to CZP 200 mg Q2W.
  Depending on PASI50 or PASI75 responses at Week 60 or a later time point, participants may have switched to CZP 400 mg Q2W or withdrew from the study.
- CZP 400 mg Q2W: CZP 400 mg Q2W through Week 14.
  Treatment received from Week 16 - 48 was based on initial treatment and response to treatment:
  * PASI50 responders at Week 16 continued to receive CZP 400 mg Q2W.
  * PASI50 non-responders at Week 16 were removed from blinded study medication and escaped to unblinded CZP 400 mg Q2W. Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study.
  * PASI50 non-responders at Week 32 or a later time point were withdrawn from the study.
  Participants who completed the Maintenance Period (with PASI50 response at Week 48) entered the OLE Period on CZP 200 mg Q2W. Week 48 completers in the escape arm continued to receive CZP 400 mg Q2W or may have switched to CZP 200 mg Q2W.
  Participants who achieved a PASI75 response during the OLE Period may have switched to CZP 200 mg Q2W.
- Placebo/Placebo Q2W: This arm consisted of participants initially randomized in the Placebo arm, who achieved a PASI75 response at Week 16 and continued to receive Placebo in the Maintenance Period (Week 16 to Week 48).
- Placebo/CZP 200 mg Q2W: This arm consisted of participants initially randomized in the Placebo arm, who achieved a PASI50 response at Week 16 but not a PASI75 response and received CZP 400 mg at Weeks 16, 18, and 20 (loading doses) followed by CZP 200 mg Q2W (starting at Week 22).
- CZP 200 mg Q2W/CZP 200 mg Q2W: This arm consisted of participants initially randomized in the CZP 200 mg Q2W arm, who achieved a PASI50 response at Week 16 and continued to receive CZP 200 mg Q2W.
- CZP 400 mg Q2W/CZP 400 mg Q2W: This arm consisted of participants initially randomized in the CZP 400 mg Q2W arm, who achieved a PASI50 response at Week 16 and continued to receive CZP 400 mg Q2W.
- Placebo/Escape CZP 400 mg Q2W: This arm consisted of participants initially randomized in the Placebo arm, who did not achieve a PASI50 response at Week 16 escaped from the blinded treatment and received unblinded CZP 400 mg Q2W, for 16 weeks. Participants who did not achieve PASI50 after 16 weeks of unblinded treatment were withdrawn from the study.
- CZP 200 mg Q2W/Escape CZP 400 mg Q2W: This arm consisted of participants initially randomized in the CZP 200 mg Q2W arm, who did not achieve a PASI50 response at Week 16 escaped from the blinded treatment and received CZP unblinded 400 mg Q2W, for 16 weeks. Participants who did not achieve PASI50 after 16 weeks of unblinded treatment were withdrawn from the study.
- CZP 400 mg Q2W/Escape CZP 400 mg Q2W: This arm consisted of participants initially randomized in the CZP 400 mg Q2W arm, who did not achieve a PASI50 response at Week 16 escaped from the blinded treatment and received unblinded CZP 400 mg Q2W, for 16 weeks. Participants who did not achieve PASI50 after 16 weeks of unblinded treatment were withdrawn from the study.
- Placebo/CZP 200 mg Q2W OLE: This arm consisted of participants who received dose-blind Placebo during the Maintenance Period, who achieved a PASI50 response at Week 48 and entered the OLE Period receiving CZP 200 mg Q2W.
- CZP 200 mg Q2W/CZP 200 mg Q2W OLE: This arm consisted of participants who received blinded CZP 200mg Q2W in the Maintenance Period, who achieved a PASI50 response at Week 48 and entered OLE on the CZP 200mg Q2W dose.
- CZP 400 mg Q2W/CZP 200 mg Q2W OLE: This arm consisted of participants who received blinded CZP 400mg Q2W in the Maintenance Period, who achieved a PASI50 response at Week 48, and entered OLE on the CZP 200mg Q2W dose.
- Escape CZP 400 mg Q2W/CZP 400 mg Q2W OLE: This arm consisted of participants who received open-label CZP 400mg Q2W in the Maintenance Period and entered OLE on the CZP 400mg Q2W dose.
Period: Initial Period (Week 0 to Week 16)
Arm/Group | Placebo Q2W | CZP 200 mg Q2W | CZP 400 mg Q2W | Placebo/Placebo Q2W | Placebo/CZP 200 mg Q2W | CZP 200 mg Q2W/CZP 200 mg Q2W | CZP 400 mg Q2W/CZP 400 mg Q2W | Placebo/Escape CZP 400 mg Q2W | CZP 200 mg Q2W/Escape CZP 400 mg Q2W | CZP 400 mg Q2W/Escape CZP 400 mg Q2W | Placebo/CZP 200 mg Q2W OLE | CZP 200 mg Q2W/CZP 200 mg Q2W OLE | CZP 400 mg Q2W/CZP 200 mg Q2W OLE | Escape CZP 400 mg Q2W/CZP 400 mg Q2W OLE
Started | 51 | 95 | 88 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Week 16 | 46 | 92 | 87 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Finished Wk16 Started Maintenance Period | 46 | 92 | 85 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 46 | 92 | 85 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse event after completing wk16 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period (Week 16 to Week 48)
Arm/Group | Placebo Q2W | CZP 200 mg Q2W | CZP 400 mg Q2W | Placebo/Placebo Q2W | Placebo/CZP 200 mg Q2W | CZP 200 mg Q2W/CZP 200 mg Q2W | CZP 400 mg Q2W/CZP 400 mg Q2W | Placebo/Escape CZP 400 mg Q2W | CZP 200 mg Q2W/Escape CZP 400 mg Q2W | CZP 400 mg Q2W/Escape CZP 400 mg Q2W | Placebo/CZP 200 mg Q2W OLE | CZP 200 mg Q2W/CZP 200 mg Q2W OLE | CZP 400 mg Q2W/CZP 200 mg Q2W OLE | Escape CZP 400 mg Q2W/CZP 400 mg Q2W OLE
Started | 0 | 0 | 0 | 3 | 5 | 74 | 77 | 38 | 18 | 8 | 0 | 0 | 0 | 0
Completed Week 48 | 0 | 0 | 0 | 3 | 5 | 71 | 70 | 33 | 13 | 7 | 0 | 0 | 0 | 0
Finished Wk48 Entered Open-label Period | 0 | 0 | 0 | 3 | 5 | 69 | 70 | 33 | 13 | 7 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 3 | 5 | 69 | 70 | 33 | 13 | 7 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 5 | 5 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Patient did not achieve PASI50 response | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Patient cannot attend visits | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No valid reason stated by patient | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not achieve PASI50 after week 48 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-label Period (Week 48 to Week 144)
Arm/Group | Placebo Q2W | CZP 200 mg Q2W | CZP 400 mg Q2W | Placebo/Placebo Q2W | Placebo/CZP 200 mg Q2W | CZP 200 mg Q2W/CZP 200 mg Q2W | CZP 400 mg Q2W/CZP 400 mg Q2W | Placebo/Escape CZP 400 mg Q2W | CZP 200 mg Q2W/Escape CZP 400 mg Q2W | CZP 400 mg Q2W/Escape CZP 400 mg Q2W | Placebo/CZP 200 mg Q2W OLE | CZP 200 mg Q2W/CZP 200 mg Q2W OLE | CZP 400 mg Q2W/CZP 200 mg Q2W OLE | Escape CZP 400 mg Q2W/CZP 400 mg Q2W OLE
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 74 | 70 | 53
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 54 | 51 | 44
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 19 | 9
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 1
Not completed — Did not achieve PASI50 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 3

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set, which consisted of all participants randomized into the study.
Arm/Group | Placebo Q2W | CZP 200 mg Q2W | CZP 400 mg Q2W | Total Title
Number analyzed (Participants) | 51 | 95 | 88 | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 90 | 86 | 221
  >=65 years | 6 | 5 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.9 (12.8) | 44.5 (13.1) | 43.6 (12.1) | 44.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 28 | 28 | 72
  Male | 35 | 67 | 60 | 162

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Achieve a Psoriasis Activity and Severity Index (PASI75) Response at Week 16
Description: The PASI75 response assessments are based on at least 75% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: At Week 16
Population: The Randomized Set included all participants randomized into the study. Missing data were handled using the Markov Chain Monte Carlo (MCMC) method for multiple imputation.
Measure: Number; unit: percentage of participants
Groups:
- Placebo Q2W (RS): Placebo sc injection Q2W.
  Treatment received from Week 16 - 48 was based on initial treatment and response to treatment:
  * PASI50 responders at Week 16, who did not achieve a PASI75 response at Week 16 received CZP 400 mg at Weeks 16, 18 and 20 (loading doses) followed by CZP 200 mg Q2W starting at Week 22.
  * PASI75 responders at Week 16 continued to receive Placebo.
  * PASI50 non-responders at Week 16 were removed from blinded study medication and escaped to unblinded CZP 400 mg Q2W. Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study.
  * PASI50 non-responders at Week 32 or a later time point were withdrawn from the study.
  Participants who completed the Maintenance Period (with PASI50 response at Week 48) entered the OLE Period on CZP 200 mg Q2W. Week 48 completers in the escape arm continued to receive CZP 400 mg Q2W or may have switched to CZP 200 mg Q2W.
  Participants formed the Randomized Set (RS).
- CZP 200 mg Q2W (RS): CZP 400 mg at Weeks 0, 2, 4, followed by CZP 200 mg Q2W from Week 6 to Week 14.
  Treatment received from Week 16 - 48 was based on initial treatment and response to treatment:
  * PASI50 responders at Week 16 continued to receive CZP 200 mg Q2W.
  * PASI50 non-responders at Week 16 were removed from blinded study medication and escaped to unblinded CZP 400 mg Q2W. Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study.
  * PASI50 non-responders at Week 32 or a later time point were withdrawn from the study.
  Participants who completed the Maintenance Period (with PASI50 response at Week 48) entered the OLE Period on CZP 200 mg Q2W.
  Week 48 completers in the escape arm continued to receive CZP 400 mg Q2W or may have switched to CZP 200 mg Q2W.
  Depending on PASI50 or PASI75 responses at Week 60 or a later time point, participants may have switched to CZP 400 mg Q2W or withdrew from the study.
  Participants formed the RS.
- CZP 400 mg Q2W (RS): CZP 400 mg Q2W through Week 14.
  Treatment received from Week 16 - 48 was based on initial treatment and response to treatment:
  * PASI50 responders at Week 16 continued to receive CZP 400 mg Q2W.
  * PASI50 non-responders at Week 16 were removed from blinded study medication and escaped to unblinded CZP 400 mg Q2W. Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study.
  * PASI50 non-responders at Week 32 or a later time point were withdrawn from the study.
  Participants who completed the Maintenance Period (with PASI50 response at Week 48) entered the OLE Period on CZP 200 mg Q2W. Week 48 completers in the escape arm continued to receive CZP 400 mg Q2W or may have switched to CZP 200 mg Q2W.
  Participants who achieved a PASI75 response during the OLE Period may have switched to CZP 200 mg Q2W.
  Participants formed the RS.
Arm/Group | Placebo Q2W (RS) | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 51 | 95 | 88
percentage of participants | 6.5 | 66.5 | 75.8
Statistical Analysis 1: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); The statistical analysis of the co-primary efficacy variables and key secondary efficacy variables accounted for multiplicity by using a fixed sequence testing procedure; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value for the primary analysis was evaluated at a 2-sided significance level of 0.025 for each CZP dose versus (vs) PBO; Estimated responder rate, odds ratios, CIs, p-values based on a logistic regression model with factors for treatment, region, prior biologic exposure; Odds Ratio (OR) = 28.962, 97.5% CI 2-sided [6.968 to 120.371]
Statistical Analysis 2: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value for the primary analysis was evaluated at a 2-sided significance level of 0.025 for each CZP dose vs PBO; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 45.660, 97.5% CI 2-sided [10.657 to 195.634]
Statistical Analysis 3: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 60.0, 95% CI 2-sided [47.92 to 72.17] — Estimate and 95% CI for difference in proportion of responders for CZP 200 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 4: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 69.3, 95% CI 2-sided [57.65 to 80.99] — Estimate and 95% CI for difference in proportion of responders for CZP 400 mg Q2W (RS) versus Placebo Q2W (RS)

2. Primary Outcome: Proportion of Subjects Who Achieve a Physician's Global Assessment (PGA) Clear or Almost Clear (With at Least 2-category Improvement) Response at Week 16
Description: The Investigator assessed the overall severity of Psoriasis (PSO) using the following 5-point scale: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W (RS) | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 51 | 95 | 88
percentage of participants | 4.2 | 47.0 | 57.9
Statistical Analysis 1: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value for the primary analysis was evaluated at a 2-sided significance level of 0.025 for each CZP dose vs PBO; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 20.116, 97.5% CI 2-sided [3.699 to 109.399]
Statistical Analysis 2: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value for the primary analysis was evaluated at a 2-sided significance level of 0.025 for each CZP dose vs PBO; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 31.143, 97.5% CI 2-sided [5.687 to 170.548]
Statistical Analysis 3: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 42.8, 95% CI 2-sided [30.70 to 54.86] — Estimate and 95% CI for difference in proportion of responders for CZP 200 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 4: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 53.6, 95% CI 2-sided [41.33 to 65.94] — Estimate and 95% CI for difference in proportion of responders for CZP 400 mg Q2W (RS) versus Placebo Q2W (RS)

3. Secondary Outcome: Proportion of Subjects Who Achieve a Psoriasis Activity and Severity Index (PASI90) Response at Week 16
Description: The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W (RS) | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 51 | 95 | 88
percentage of participants | 0.4 | 35.8 | 43.6
Statistical Analysis 1: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value for this analysis as used in the fixed sequence testing procedure was evaluated at a 2-sided significance level of 0.025 for each CZP dose vs PBO; Estimated responder rate, odds ratios, CIs, p-values based on a logistic regression model with factors for treatment,region, prior biologic exposure; Odds Ratio (OR) = 36.668, 97.5% CI 2-sided [5.717 to 235.193]
Statistical Analysis 2: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 50.606, 97.5% CI 2-sided [7.880 to 324.988]
Statistical Analysis 3: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 35.4, 95% CI 2-sided [20.85 to 49.87] — Estimate and 95% CI for difference in proportion of responders for CZP 200 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 4: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 43.1, 95% CI 2-sided [27.56 to 58.71] — Estimate and 95% CI for difference in proportion of responders for CZP 400 mg Q2W (RS) versus Placebo Q2W (RS)

4. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a subject-reported questionnaire designed for use in adult participants with PSO. The DLQI is a skin disease-specific questionnaire aimed at the evaluation of how symptoms and treatment affect patients' health related quality of life (HRQoL). This instrument asks participants about symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. It has been shown to be valid and reproducible in PSO patients. The DLQI score ranges from 0 to 30 with higher scores indicating lower HRQoL. A higher than of equal to (>=) 4-point change in the DLQI score (DLQI response) has been reported to be meaningful for the patient (within-patient minimal important difference Basra et al, 2015) a DLQI absolute score of lower than or equal to (=<) 1 indicates DLQI remission (i.e., no or small impact of the disease on HRQoL).
Time Frame: At Week 16
Population: The Randomized Set included all participants randomized into the study. Missing data were handled using the last observation carried forward (LOCF) method for the DLQI.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo Q2W (RS) | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 51 | 95 | 88
Scores on a scale | -3.3 (0.80) | -9.3 (0.58) | -10.2 (0.60)
Statistical Analysis 1: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — P-value obtained for each treatment group comparison tested at a significance level of 0.025 in the fixed sequence testing procedure; ANCOVA model of change from Baseline DLQI score with treatment group, region, prior biologic exposure as factors; Baseline DLQI score as a covariate; Adjusted Mean Treatment Differences = -6.00, 97.5% CI 2-sided [-8.18 to -3.81]
Statistical Analysis 2: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]; Ajusted Mean Treatment Differences = -6.84, 97.5% CI 2-sided [-9.05 to -4.62]

5. Secondary Outcome: Proportion of Subjects Who Achieve a Physician's Global Assessment (PGA) Clear or Almost Clear (With at Least 2-category Improvement) Response at Week 48
Description: The Investigator assessed the overall severity of Psoriasis (PSO) using the following 5-point scale: 0= clear, 1= almost clear, 2= mild, 3= moderate, 4= severe.
Time Frame: At Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 95 | 88
percentage of participants | 52.7 [41.99 to 63.32] | 69.5 [59.24 to 79.77]

6. Secondary Outcome: Proportion of Subjects Who Achieve a Psoriasis Activity and Severity Index (PASI75) Response at Week 48
Description: as for outcome 1
Time Frame: At Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 95 | 88
percentage of participants | 67.2 [57.09 to 77.39] | 87.1 [79.81 to 94.45]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Baseline (Week 0) until the Post Study Safety Follow-up Visit (Week 152).
Description: Participants randomized to PBO switched to CZP 200mg Q2W or CZP 400mg Q2W at Week 16. Participants randomized to CZP were exposed for up to 144 weeks, leading to a significantly lower exposure in the PBO than CZP arm. Considering the imbalance of such comparison, AEs reported while participants were on PBO are not included in this summary.
Groups:
- CZP 200 mg Q2W (TCS): This arm consisted of all participants who received CZP 200 mg at any time during the study.
- CZP 400 mg Q2W (TCS): This arm consisted of all participants who received CZP 400 mg at any time during the study.
Arm/Group | CZP 200 mg Q2W (TCS) | CZP 400 mg Q2W (TCS)
All-Cause Mortality (participants affected / at risk) | 1/188 | 1/167
Serious Adverse Events (participants affected / at risk) | 14/188 | 19/167
Other Adverse Events (participants affected / at risk) | 95/188 | 85/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CZP 200 mg Q2W (TCS) (N=188) | CZP 400 mg Q2W (TCS) (N=167)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Blepharochalasis (Eye disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactoid reaction (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Borrelia infection (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CZP 200 mg Q2W (TCS) (N=188) | CZP 400 mg Q2W (TCS) (N=167)
Nasopharyngitis (Infections and infestations) | 54 (86) | 51 (95)
Upper respiratory tract infection (Infections and infestations) | 21 (28) | 26 (42)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (16) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 11 (12)
Headache (Nervous system disorders) | 9 (18) | 14 (41)
Psoriasis (Skin and subcutaneous tissue disorders) | 9 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days